CLINICAL TRIAL: NCT01165372
Title: Clinical Investigation of In-vivo Susceptibility of P. Falciparum to Artesunate in Phuoc Long Hospital, Binh Phuoc Province, Vietnam
Brief Title: Study of Malaria Treatment at Phuoc Long Hospital, Binh Phuoc Province, Vietnam
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oxford University Clinical Research Unit, Vietnam (Other)
Collaborators: World Health Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 02MA
Record Dates: First submitted 2010-07-15; First posted 2010-07-19 (Estimated); Last update posted 2011-09-15 (Estimated); Status verified 2011-09

CONDITIONS: Malaria
Keywords: Malaria; Drug resistance
MeSH Terms: conditions — Malaria | interventions — Artesunate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Artesunate 2mg (Experimental): People with uncomplicated malaria who meet the study inclusion criteria will be enrolled, screened, randomized and treated on site with artesunate 2mg/kg/day for 3 days and followed by DHA-PPQ treatment at doses according to National guidelines for 3 days.
  Interventions: Drug: Artesunate or dihydroartemisinin-piperaquine
- Artesunate 4mg (Experimental): People with uncomplicated malaria who meet the study inclusion criteria will be enrolled, screened, randomized and treated on site with artesunate 4mg/kg/day for 3 days and followed by DHA-PPQ treatment at doses according to National guidelines for 3 days.
  Interventions: Drug: Artesunate or dihydroartemisinin-piperaquine
- DHA-piperaquine (Experimental): People with uncomplicated malaria who meet the study inclusion criteria will be enrolled, screened, randomized and treated on site with dihydroartemisinin-piperaquine once daily according to weight for 3 days.
  Interventions: Drug: Artesunate or dihydroartemisinin-piperaquine

INTERVENTIONS:
Drug: Artesunate or dihydroartemisinin-piperaquine — artesunate 2mg/kg/day, artesunate 4mg/kg/day or dihydroartemisinin-piperaquine once daily

SUMMARY:
Background: There are worrying signs from Western Cambodia that parasitological responses to artesunate containing treatment regimens for uncomplicated falciparum malaria are slower than elsewhere in the world. Delayed parasite clearance and unusually high failure rates with artesunate-mefloquine have been reported. These antimalarials are central to current treatment strategies and spread of significant resistance outside this area would be a global disaster. Radical containment measures are needed. In this context there is an urgent need to proceed quickly to investigate whether there is any evidence of resistance to artemisinin derivatives in Vietnam.

Objective: The primary objective is to assess the slope of the decline in the log parasitemia-time curve in patients treated with artesunate 2mg/kg/day, artesunate 4mg/kg/day or dihydroartemisinin-piperaquine once daily, and to compare the results of this study to the pharmacokinetic results and to the recent data from patients in Cambodia and Thailand treated with equivalent therapies.

Methods: The trial will be conducted in Phuoc Long Hospital, Binh Phuoc Province, Vietnam. The participants will be febrile patients (aged > 10 years) with slide confirmed uncomplicated P. falciparum infection. Patients will be treated with either artesunate 2mg/kg/day, artesunate 4mg/kg/day or dihydroartemisinin-piperaquine once daily for 3 days. Patients on artesunate therapy arms will then receive 3 days of treatment with dihydroartemisinin-piperaquine with dosages according to the national guidelines. Clinical and parasitological parameters will be monitored over a 42-day follow-up period. The pharmacokinetic characteristics of artesunate and dihydroartemisinin will be assessed by using a population pharmacokinetic modeling.

DETAILED DESCRIPTION:
This surveillance study is a three-arm prospective evaluation of the efficacy of artesunate and dihydroartemisinin-piperaquine in acute uncomplicated falciparum malaria. This will be an evaluation of the slope of the decline in the log parasitemia-time curve, parasite clearance times in patients randomized to one of two different doses of oral artesunate or dihydroartemisinin-piperaquine. People with uncomplicated malaria who meet the study inclusion criteria will be enrolled, screened, randomized and treated on site with either artesunate 2mg/kg/day, artesunate 4mg/kg/day or dihydroartemisinin-piperaquine once daily according to weight for 3 days. The artesunate arms will immediately follow with dihydroartemisinin-piperaquine therapy for 3 days (study days 3 - 6) at the dose defined by national guidelines. Patients on all three arms will be monitored for 42 days. The follow-up will consist of a fixed schedule of check-up visits and corresponding clinical and laboratory examinations. PCR analysis will be used to distinguish between true recrudescence due to treatment failure and reinfection.

ELIGIBILITY:
Inclusion Criteria:

* male and aged > 10 years OR;
* female patients > 10 and <12 years old, provided they have not reached menarche
* mono-infection with P. falciparum detected by microscopy;
* parasitaemia of 10,000 - 100,000/µl asexual forms;
* presence of axillary or tympanic temperature ≥ 37.5 °C or history of fever during the past 24 h;
* ability to swallow oral medication;
* ability and willingness to comply with the study protocol for the duration of the study and to comply with the study visit schedule;
* informed consent/assent.

Exclusion Criteria:

* presence of general danger signs or severe falciparum malaria according to the definitions of WHO;
* mixed or mono-infection with another Plasmodium species detected by microscopy;
* presence of severe malnutrition (defined as a child whose growth standard is below -3 z-score, has symmetrical oedema involving at least the feet or has a mid-upper arm circumference < 110 mm);
* presence of febrile conditions due to diseases other than malaria (e.g. measles, acute lower respiratory tract infection, severe diarrhoea with dehydration) or other known underlying chronic or severe diseases (e.g. cardiac, renal and hepatic diseases, HIV/AIDS);
* regular medication, which may interfere with antimalarial pharmacokinetics;
* treatment with antimalarial drugs in the previous 48 hours;
* history of hypersensitivity reactions or contraindications to any of the medicine(s) being tested or used as alternative treatment(s);
* splenectomy.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2010-08; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Slope of the decline in the log parasitemia-time curve relative to historical data | 03 days

SECONDARY OUTCOMES:
Clearance rate assessed from the fitted slope of the log-linear parasite curves | 72 hours
Proportion of patients who have a parasite clearance time >72 hours after initiation of each treatment | 72 hours
Parasitological efficacy of the three treatment arms | Over 72 hours and during follow-up treatment over a total follow-up period of 42 days
Relative proportion of patients treated with artesunate 2mg/kg/day versus artesunate 4mg/kg/day versus dihydroartemisinin-piperaquine once daily | 03 days
  Patients who result as early treatment failures, late clinical failures, late parasitological failures or adequate clinical and parasitological response as indicators of efficacy
Recrudescence and new infection rate defined by polymerase chain reaction (PCR) analysis between treatment arms | 42 days
Number of adverse events in each treatment arm | After initiation and during follow-up treatment over a total follow-up period of 42 days.
Assess the pharmacokinetic characteristics of artesunate and dihydroartemisinin-piperaquine by using population pharmacokinetic modeling | 03 days and upon relapse
Characterize different genetic patterns from different resistant strains | 03 days

CONTACTS AND LOCATIONS:
Overall Officials: Hien T Tran, MD, PhD, Principal Investigator — Oxford University Clinical Research Unit, Vietnam
Locations (1):
- Phuoc Long Hospital, Dong Xoai, Binh Phuoc, Vietnam

REFERENCES:
- See also: Related Info — http://www.oucru.org